CLINICAL TRIAL: NCT06987981
Title: A Randomized, Open Label, Two-arm Study: Evaluation of Burn Wound and Scar Healing Time in Paediatric Burn Patients Using Chitosan-Based vs. Silver-Based Dressings
Brief Title: Comparing How Burn Wounds and Scars Heal in Children Using Chitosan and Silver Dressings
Acronym: CHITAG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Miloš Potkonjak (Other)
Collaborators: General Hospital of Novo mesto (Other)
Responsible Party: Sponsor-Investigator, Miloš Potkonjak, MD, surgeon, General Hospital of Novo mesto
Organization: General Hospital of Novo mesto (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHITAG-25-01
Record Dates: First submitted 2025-05-09; First posted 2025-05-23 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-05

CONDITIONS: Burns Degree Second; Pediatric
Keywords: Chitosan-based dressing; Silver-based dressing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chitosan group (Active Comparator): Chitosan group - using chitosan-based dressing for wound and scar treatment
  Interventions: Device: Chitosan-based dressing
- Ag group (Active Comparator): Ag group - using silver-based dressing, followed by a cosmetic lotion
  Interventions: Device: Silver-based dressing

INTERVENTIONS:
Device: Chitosan-based dressing — Chitosan-based dressing for wound and scar treatment will be used (e.g. ChitoCare® medical Wound Healing Gel)
  Arms: Chitosan group
Device: Silver-based dressing — Silver-based dressing (e.g. AQUACEL® Ag), followed by a cosmetic lotion (e.g.: Bepanthol® DERMA) will be used
  Arms: Ag group

SUMMARY:
Burns are among the most common types of trauma worldwide, ranking fourth after traffic accidents, falls, and violence, and account for an estimated 265,000 deaths annually (WHO). Most burn injuries result from heat exposure, though other causes include friction, chemicals, and electricity. Effective burn treatment aims to promote wound healing by supporting tissue regeneration and maintaining optimal conditions such as moisture, oxygenation, and low bacterial load.

In Slovenia and across Europe, silver-based dressings are commonly used for burn care. While they are known to support wound healing, their effectiveness in reducing scar formation remains unclear. Chitosan-based hydrogels, by contrast, offer promising benefits due to their natural biocompatibility, antibacterial action, and support for tissue repair, though clinical data are still limited.

This study aims to compare the effectiveness of chitosan-based and silver-based dressings in burn wound healing, focusing on healing time, scar formation, cost-efficiency, and patient experience. Scar outcomes will be assessed using the validated POSAS (Patient and Observer Scar Assessment Scale).

ELIGIBILITY:
Inclusion Criteria:

1. Age between 6 months and 17 years old
2. Having a first or second-degree superficial burn that does not require excision and grafting
3. Patients with a burn of less than 20% of the total body surface area (TBSA)
4. Admission within 72 hours of burn injury
5. First line of therapy is Burnshield® Dressing for the first 48 hours
6. Clean non-infected wound as diagnosed by the attending physician
7. Informed consent of the patient or caregiver

Exclusion Criteria:

1. Causes other than contact burn, flame or scald injuries (i.e., electrical, chemical or frostbite)
2. Diabetes mellitus
3. Significant cardiac, pulmonary, or renal insufficiency
4. Severe hematologic disease, malignancy, hypo-immunity
5. Wounds noted to be contaminated or infected
6. Systemic inflammatory response syndrome (SIRS) or sepsis
7. Moderate or severe respiratory tract or lungs burn injuries
8. Previous treatment efforts such as previous debridement, silver sulfadiazine ointment or other topical agents (e.g.: oil, toothpaste, betadine, rivano)
9. Being pregnant or breastfeeding
10. Known sensitivity or allergy to one of the dressings or its components.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Wound Healing Time | Up to 21 days
  To evaluate and compare the wound healing time, measured as the number of days required for complete healing of the study wound, between the treatment groups.

SECONDARY OUTCOMES:
Wound Healing Rate | 7, 14, and 21 days
  To evaluate and compare the wound healing rate, calculated as the ratio of the healed wound area to the initial wound area, at 7, 14, and 21 days of treatment
Complete Wound Healing Rate | 21 days
  To assess and compare the percentage of patients achieving complete wound healing within 21 days of treatment
Scar Outcomes | 1, 3, and 6 months
  To evaluate and compare scar outcomes of treated burn wounds using a validated scar assessment tool Patient and Observer Scar Assessment Scale (POSAS) at 1 month, 3 months, and 6 months after injury. POSAS measures subjective assessment on a 1-10 scale from normal skin to worst scar imaginable across 6 metrics (surface area, vascularity, pigmentation, thickness, pliability and relief). The lowest sum score, reflecting normal skin, is 6 and the highest score, reflecting the worst imaginable scar, is 60.
Cost-effectiveness | 21 days
  To assess the cost-effectiveness of the treatment (e.g.: number of dressing changes required, number of hospital visits, costs of additional therapies related to wound healing (e.g., pain relievers)), at 21 days of treatment.
Professional Experience | 0, 7, 14, and 21 days
  Medical staff will complete a survey consisting of 4 items evaluating their experience with the selected therapy. The survey includes questions addressing the complexity of the wound care therapy-such as its application, removal, and time requirements-as well as overall satisfaction. Responses will be collected using a combination of Yes/No/Not sure options and a Visual Analogue Scale (VAS), where 0 indicates "Not at all" and 5 indicates "Very much."
Patient Experience | 0, 7, 14 and 21 days, and 1, 3, and 6 months
  Patients will complete a survey consisting of 4 to 7 items evaluating their experience with the burn wound or scar treatment procedure. The survey includes questions related to patient satisfaction, which are a combination of Yes/No/Not sure responses and a visual analogue scale (VAS), where 0 represents "Not at all" and 5 represents "Very much." Additionally, questions addressing the patient's response to treatment use face scale items scored from 0 to 10, assessing symptoms such as pain, heat, itching, and irritation. A score of 0 corresponds to "Not at all," while a score of 10 indicates "Very much," with higher scores reflecting greater intensity of the respective symptom.
Adverse Events | up to 21 days
  To assess the proportion of patients who experience adverse events associated with the dressing, from the time of admission up to 21 days of treatment.
Rate of Infection | up to 1 month
  To evaluate the rate of infection in burn wounds, defined as the number of infected wounds divided by the total number of burn wounds, assessed at each study visit up to 1 month of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Miloš Potkonjak, MD, surgeon, Principal Investigator — General Hospital of Novo mesto
Locations (1):
- General Hospital Novo mesto, Novo Mesto, Slovenia

IPD SHARING:
Plan to Share IPD: No
As an Institution operating under the jurisdiction of the European Union, we are subject to the General Data Protection Regulation (GDPR), which imposes strict requirements on the processing and sharing of personal data, including health-related information. IPD from clinical trials is considered sensitive personal data under GDPR.
  Even when data is anonymized or pseudonymized, sharing IPD with third parties-especially outside the EU-requires careful assessment of data protection safeguards, appropriate legal basis, and in some cases, additional participant consent. Unless all conditions for lawful data transfer and processing are met, including compliance with GDPR Articles 44-50 concerning international data transfers, we are not permitted to share IPD.
  For this reason, and in order to ensure full compliance with EU data protection regulations and to protect the privacy and rights of our study participants, we are currently unable to share individual-level clinical trial data.